CLINICAL TRIAL: NCT01015755
Title: Palliation of Thirst in ICU Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Kathleen Puntillo, Professor of Nursing, Emeritus, University of California, San Francisco
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01NR011825-01 (NIH)
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Thirst
Keywords: thirst palliation and intensive care unit; thirst intensity and distress; predictors of thirst

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- thirst intervention (Experimental)
  Interventions: Behavioral: combined therapy treatment

INTERVENTIONS:
Behavioral: combined therapy treatment — mouth care

SUMMARY:
Patients in Intensive Care Units are often extremely thirsty due to their medicines, illness, treatments or medicines that they receive. This study will test whether patients who receive a easy to implement intervention for thirst will have greater relief from thirst than a group of patients who do not receive the intervention. The study will also identify the most important factors that make ICU patients thirsty so that future research studies can test how to relieve those factors and/or make interventions for thirst more readily available.

DETAILED DESCRIPTION:
This study will test the efficacy of an innovative, inexpensive, resource-efficient treatment for thirst -- one of the most pervasive, intense, unrecognized, and under-treated symptoms suffered by critically ill patients in Intensive Care Units (ICUs). The first aim of this single-blinded, randomized clinical trial is to test a non-pharmacologic intervention for thirst in ICU patients. The intervention is a combination therapy treatment (CTT) for thirst that includes the use of sterile water mouth sprays, sterile water swabs, and menthol-based lip and tongue moisturizer. The second aim of the study is to examine demographic, environmental, and health and illness factors that increase an ICU patient's risk profile for thirst. Aim #1 hypotheses: (1) Thirst intensity and distress will decrease significantly in ICU patients who receive a CTT for thirst compared to those who receive research team observation. (2) Subjective (e.g., dry mouth) and objective (e.g., cracked lips) thirst-related characteristics will decrease significantly in ICU patients who receive a CCT for thirst compared to those who receive research team observation. Aim #2 hypotheses: (1) A significant association will be found between presence of thirst and certain risk factors for thirst, e.g., serum osmolality, hydration status, and administration of certain medications, e.g., opioids. (2) A significant association will be found between the intensity of thirst and certain risk factors for thirst, e.g., serum osmolality, hydration status, and administration of certain medications, e.g., opioids.

The sample will be 245 ICU patients in one Experimental and two Control groups. Those with thirst will be randomized to either the Experimental or the Control 1 group. The Experimental group will receive the CTT; the Control 1 group will receive research team observation. The Control 2 group patients who reported no thirst will be compared to the Control 1 group on characteristics associated with the presence and intensity of thirst.

Multilevel linear regression models will be employed to test the difference in the linear change trajectories between the treatment and control groups. Multiple logistic regression analysis and multiple linear regression analysis will be used to determine association of risk factors with the presence and intensity of thirst, respectively.

Results will contribute empirical data needed to stimulate a far overdue nursing practice change for the treatment of thirst in ICUs. Results will also identify a risk profile for thirst that will be an important target for future research of thirst in ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* must be able to self-report thirst intensity or distress

Exclusion Criteria:

* unable to self-report thirst
* comatose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2010-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Thirst intensity | after thirst intervention

SECONDARY OUTCOMES:
Thirst distress | after thirst intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen A Puntillo, RN, DNSc, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Puntillo K, Arai SR, Cooper BA, Stotts NA, Nelson JE. A randomized clinical trial of an intervention to relieve thirst and dry mouth in intensive care unit patients. Intensive Care Med. 2014 Sep;40(9):1295-302. doi: 10.1007/s00134-014-3339-z. Epub 2014 Jun 4. PMID 24894026